CLINICAL TRIAL: NCT05101369
Title: An Open-Label Study Assessing the Mass Balance, Pharmacokinetics, and Metabolite Profiles of a Single Oral Dose of [14C]-INCB086550
Brief Title: A Study Assessing the Mass Balance, Pharmacokinetics, and Metabolite Profiles of a Single Oral Dose of [14C]-INCB086550
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 86550-106; 2020-005879-12 (EudraCT Number)
Record Dates: First submitted 2021-10-06; First posted 2021-11-01 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers; male only

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INCB086550 (Experimental): Participants will be administered INCB086550 orally, followed approximately 10 minutes later by an oral dose solution of radio labeled INCB086550.
  Interventions: Drug: INCB086550

INTERVENTIONS:
Drug: INCB086550 — INCB086550 will be administered orally, followed approximately 10 minutes later by an oral dose solution of radio labeled INCB086550.

SUMMARY:
To evaluate the absorption, metabolism, and excretion of 86550-106 in healthy males.

DETAILED DESCRIPTION:
The purpose of this study is to determine the absorption, metabolism, and excretion of a single oral dose of 400 mg (4x100 mg tablets) of INCB086550 followed by an oral dose solution of approximately 100 μCi (3.7 MBq) [14C]-INCB086550 and to characterize and determine the metabolites present in plasma, urine, and, where possible, feces in healthy male participants .

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Male healthy adult participants aged 35 to 55 years, inclusive, at the time of screening.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, at the time of screening.
* No clinically significant findings in screening evaluations (clinical, laboratory, vital signs, and ECG).
* Ability to swallow and retain oral medication.
* Willingness to avoid fathering children based on the criteria below. a. Male participants with reproductive potential must agree to take appropriate precautions to avoid fathering children from screening through 90 days (a spermatogenesis cycle) after the dose of study drug and must refrain from donating sperm during this period. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.

Exclusion Criteria:

History of clinically significant respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease.

* History of cardiovascular, cerebrovascular, peripheral vascular, or thrombotic disease or uncontrolled hypertension (systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mmHg at screening, confirmed by repeat testing).
* History of rheumatologic/autoimmune disorders, except for minor eczema and rosacea.
* Resting pulse < 40 bpm or > 100 bpm, confirmed by repeat testing at screening.
* History or presence of an abnormal ECG at screening or predose on Day 1 that, in the investigator's opinion, is clinically significant. QTcF interval > 450 milliseconds, QRS interval > 120 milliseconds, and PR interval > 220 milliseconds.
* Presence of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn's disease or chronic pancreatitis). Hemoglobin, WBC, platelet, or absolute neutrophil count that is out of the laboratory's range unless considered clinically insignificant by the investigator at screening or check-in.
* Hepatic transaminases (ALT and AST), ALP, or total bilirubin > 1.25 × the laboratory-defined ULN at screening or check-in, confirmed by repeat testing (except participants with Gilbert's disease, for which total bilirubin must be ≤ 2.0 × ULN).
* History of malignancy within 5 years of screening, with the exception of cured basal cell or squamous cell carcinoma of the skin.
* Current or recent (within 6 months of screening) clinically significant gastrointestinal disease or surgery (including cholecystectomy, excluding appendectomy) that could affect the absorption of study drug.
* Any major surgery within 6 months of screening.
* Donation of blood to a blood bank or in a clinical study (except a screening visit) within 3 months of screening (within 2 weeks for plasma donation).
* Blood transfusion within 4 weeks of check-in.
* Chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment (includes any history of tuberculosis).
* Positive test for HBV, HCV, or HIV. Participants whose results are compatible with prior immunization or immunity due to infection for HBV may be included at the discretion of the investigator.
* History of alcohol dependency within 3 years of screening.
* Consumption of alcohol 72 hours before check-in (Day -1) until CRU discharge.
* Positive breath test for alcohol or positive urine screen for drugs of abuse (confirmed by repeat) at screening or check-in that are not otherwise explained by permitted concomitant medications.
* Current treatment or treatment within 90 days or 5 half-lives (whichever is longer) prior to dosing in this study with another investigational medication or current enrollment in another investigational drug study.
* Participated in any clinical study involving a radiolabeled investigational product within 12 months prior to check-in.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) prior to dosing in this study with any medications known to be an inducer or inhibitor of CYP3A4, P-gp, or BCRP (refer to the Drug Interaction Database Program [University of Washington School of Pharmacy 2002] for prohibited drugs).
* Consumption of Seville oranges, grapefruit, pomelos, exotic citrus fruits, grapefruit hybrids, or any fruit juices (including but not limited to juices containing Seville orange, grapefruit, pomelo, exotic citrus fruits, or grapefruit hybrids) within 72 hours prior to dosing until CRU discharge.
* Consumption of poppy seeds within 7 days prior to screening and check-in. Consumption of caffeine- or xanthine-containing products (eg, coffee, tea, cola drinks, and chocolate) for 72 hours prior to dosing until CRU discharge.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator.
* Known hypersensitivity or severe reaction to INCB086550 or any excipients of INCB086550 (refer to the IB).
* Inability to undergo venipuncture or tolerate venous access.
* Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations, in the opinion of the investigator.
* History of tobacco- or nicotine-containing product use within 1 month of screening.

Consumption of tobacco- or nicotine-containing products 72 hours before check-in (Day -1) until CRU discharge is not permitted.

* Participation in strenuous exercise from 7 days before check-in until CRU discharge.
* Use of prescription drugs within 14 days of study drug administration or nonprescription medications/products (including vitamins, minerals, and phytotherapeutic, herbal, or plant-derived preparations) within 7 days prior to study drug administration and during the study. However, paracetamol up to 1000 mg Q24H and ibuprofen up to 600 mg Q24H are permitted.
* Use or intention to use any COVID-19 vaccine within 30 days prior to Day 1 and through CRU discharge or ET.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* eGFR < 90 mL/min/1.73 m2 based on the site's preferred formula at screening, check-in,or both.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male participants meeting all of the inclusion and none of the exclusion criteria.
Enrollment: 7 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Total recovery of radioactivity from urine and feces. | Approximately 2 weeks
  To determine the route of elimination and mass balance of [14C]-INCB086550 following administration of a single oral dose of 400 mg of INCB086550 followed by an oral dose solution of approximately 100 μCi (3.7 MBq) [14C]-INCB086550.
Percentage of total radioactive dose in Plasma, Urinary and Fecal Excretion | Up to approximately 2 months
  To characterize the metabolic profile and identify circulating and excreted metabolites of INCB086550 following administration of a single oral dose of 400 mg of INCB086550 followed by an oral dose solution of approximately 100 μCi (3.7 MBq) [14C]-INCB086550 using liquid chromatography with mass spectral detection.

SECONDARY OUTCOMES:
PK for plasma INCB086550: Cmax | Pre dose and Post dose on Day 1, Post dose Day 2, post dose Day 3, post dose Day 4, post dose Day 5
  Maximum Observed Plasma Concentration of INCB086550 to evaluate the PK of total radioactivity and parent compound following administration of a single oral dose of 400 mg of INCB086550 followed by an oral dose solution of approximately 100 μCi (3.7 MBq) [14C]-INCB086550.
PK for plasma INCB086550: tmax | Pre dose and Post dose on Day 1, Post dose Day 2, post dose Day 3, post dose Day 4, post dose Day 5
  Time to reach maximum (peak) Plasma concentration of INCB086550
PK for plasma INCB086550: AUC0-t | Pre dose and Post dose on Day 1, Post dose Day 2, post dose Day 3, post dose Day 4, post dose Day 5
  Area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration of INCB086550
PK for plasma INCB086550: AUC0-∞ | Pre dose and Post dose on Day 1, Post dose Day 2, post dose Day 3, post dose Day 4, post dose Day 5
  area under the single-dose plasma concentration-time curve from Hour 0 to infinity of INCB086550
PK for plasma INCB086550: t½ | Pre dose and Post dose on Day 1, Post dose Day 2, post dose Day 3, post dose Day 4, post dose Day 5
  AUC to the end of dosing period of INCB086550
PK for plasma INCB086550: λz | Pre dose and Post dose on Day 1, Post dose Day 2, post dose Day 3, post dose Day 4, post dose Day 5
  Terminal elimination rate constant of INCB086550
PK for plasma INCB086550: CL/F | Pre dose and Post dose on Day 1, Post dose Day 2, post dose Day 3, post dose Day 4, post dose Day 5
  Oral dose clearance of INCB086550
PK for plasma INCB086550: Vz/F | Pre dose and Post dose on Day 1, Post dose Day 2, post dose Day 3, post dose Day 4, post dose Day 5
  Apparent oral dose volume of distribution of INCB086550
PK for Urine INCB086550: Ae | Pre dose and Post dose daily up to day 11, until study discharge
  Cumulative amount of unchanged drug excreted into the urine. Urine will be collected for the following intervals relative to study treatment administration: -12 to 0 hours (predose void [spot sample] only) and 0 to 6, 6 to 12, and 12 to 24 hours postdose and continuing in 24-hour intervals until discharge.
PK for urine INCB086550: CLR | Pre dose and Post dose daily up to day 11, until study discharge
  Renal clearance of the drug from plasma.
PK for Urine INCB086550: fe | Pre dose and Post dose daily up to day 11, until study discharge
  Fraction of the intravenously administered drug excreted into the urine
PK for whole blood and plasma total radioactivity: Cmax | Pre dose and poste dose Day 1, post dose Days 2, 3, 4, 5 and Days 6-11 as needed until study discharge
  Maximum Observed Plasma Concentration
PK for whole blood and plasma total radioactivity: tmax | Pre dose and post dose Day 1, post dose Days 2, 3, 4, 5 and Days 6-11 as needed until study discharge
  Time to reach maximum (peak)
PK for whole blood and plasma total radioactivity: t½ | Pre dose and post dose Day 1, post dose Days 2, 3, 4, 5 and Days 6-11 as needed until study discharge
  To evaluate the PK of total radioactivity and parent compound following administration of a single oral dose of 400 mg of INCB086550 followed by an oral dose solution of approximately 100 μCi (3.7 MBq) [14C]-INCB086550.
PK for whole blood and plasma total radioactivity: AUC0-t | Pre dose and post dose Day 1, post dose Days 2, 3, 4, 5 and Days 6-11 as needed until study discharge
  Area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration of INCB086550
PK for whole blood and plasma total radioactivity: AUC0-∞ | Pre dose and post dose Day 1, post dose Days 2, 3, 4, 5 and Days 6-11 as needed until study discharge
  To evaluate the PK of total radioactivity and parent compound following administration of a single oral dose of 400 mg of INCB086550 followed by an oral dose solution of approximately 100 μCi (3.7 MBq) [14C]-INCB086550.
Incidence of AEs, ECGs, vital signs, and clinical laboratory evaluation. | up to approximately 3 months
  To evaluate the safety of a single oral dose of 400 mg of INCB086550 followed by an oral dose solution of approximately 100 μCi (3.7 MBq) [14C]-INCB086550.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Getsy, Study Director — Incyte Corporation
Locations (1):
- Covance Leeds Cru, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No